CLINICAL TRIAL: NCT03148366
Title: Comparison of the Efficacy of Levofloxacin-based Sequential Therapy and Bismuth Quadruple Therapy in the Second Line and Third Line Therapy for Helicobacter Pylori Infection- A Multi-center Randomized Trial
Brief Title: Comparison of the Levofloxacin Sequential Therapy and Quadruple Therapy in Second Line Treatment for HP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 201410001MINC
Record Dates: First submitted 2015-01-30; First posted 2017-05-11 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2017-03

CONDITIONS: Helicobacter
Keywords: Self Efficacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levofloxacin based sequential therapy (Experimental): Levofloxacin based sequential therapy
  : sequential therapy containing levofloxacin for 14 days D1-D7: (esomeprazole 40mg bid + amoxicillin 1gm bid) for 7 days D8-D14: (esomeprazole 40mg bid + levofloxacin 250mg bid + metronidazole 500mg bid) for another 7 days
  Interventions: Drug: Levofloxacin based sequential therapy
- bismuth quadruple therapy (BQ) (Active Comparator): bismuth quadruple therapy for 10 days (BQ) D1-D10: (esomeprazole 40mg bid + Dibismuth trioxide 120mg qid + metronidazole 500mg tid + tetracycline 500mg qid) for 10 days
  Interventions: Drug: bismuth quadruple therapy for 10 days (BQ)

INTERVENTIONS:
Drug: Levofloxacin based sequential therapy — D1-D7: (esomeprazole 40mg bid + amoxicillin 1gm bid) for 7 days D8-D14: (esomeprazole 40mg bid + levofloxacin 250mg bid + metronidazole 500mg bid) for another 7 days
  Arms: Levofloxacin based sequential therapy
Drug: bismuth quadruple therapy for 10 days (BQ) — D1-D10: (esomeprazole 40mg bid + Dibismuth trioxide 120mg qid + metronidazole 500mg tid + tetracycline 500mg qid) for 10 days
  Arms: bismuth quadruple therapy (BQ)

SUMMARY:
Objectives: Eradication of H. pylori infection could reduce the occurence or recurrence of gastric cancer and peptic ulcer diseases. However, it was estimated that 15-20% of patients would fail from first line standard eradication therapy and need second line rescue therapy. About 15-30% of patient would fail from second line therapy. Bismuth quadruple therapy and triple therapy containing levofloxacin are currently the recommended rescue therapies in the second line and third line treatment. Recently, our pilot study showed that modified sequential therapy containing levofloxacin achieved high eradication rate (95%) in the second line therapy. The regimen includes a PPI plus amoxicillin for 5-7 days, followed by a PPI plus levofloxacin and metronidazole for another 5-7 days. However, whether this modified sequential therapy containing levofloxacin is more effective than bismuth quadruple therapy in the second line and third line treatment remains unknown. Besides, the impact of these regimens on the antibiotic resistance , microbiota of gut flora, and metabolic factors remains unknown.

Aims: Therefore, the investigators aimed to

1. compare the eradication rates and long term re-infection rates of sequential therapy containing levofloxacin for 14 days versus bismuth quadruple therapy for 10 days in the second line and third line treatment
2. assess the impact of antibiotic resistance and CYP2C19 polymorphism on the eradication rate of these regimens
3. assess the impact of these eradication regimens on the antibiotic resistance and microbiota of the gut flora
4. assess the impact of eradication therapy on the metabolic factors

DETAILED DESCRIPTION:
Methods:

This will be a multi-center, open labeled, randomized comparative trial with cross-over design Patients: Participants with refractory H. pylori infection after one eradication therapy

Testing for H. pylori infection Before Second Line Treatment : Any two positive of CLO test, histology, and culture or a positive UBT will be considered as H. pylori infected

After Second Line Treatment: C13-UBT will be used to assess the existence of H. pylori 6-8 weeks after first line therapy.

Long term reinfection: C13-UBT will be used to assess the recurrence of H. pylori 1 year after eradication therapy

Interventions:

Second line therapy: eligible patients will be randomized into one of the two groups Group (A): sequential therapy containing levofloxacin for 14 days (EAML) D1-D7: (esomeprazole 40mg bid + amoxicillin 1gm bid) for 7 days D8-D14: (esomeprazole 40mg bid + levofloxacin 250mg bid + metronidazole 500mg bid) for another 7 days

Group (B): bismuth quadruple therapy for 10 days (BQ) D1-D10: (esomeprazole 40mg bid + Dibismuth trioxide 120mg qid + metronidazole 500mg tid + tetracycline 500mg qid) for 10 days

Third line therapy: patients who fail from second line treatment will be rescue with the following treatment Group (A) Patient who fail from levofloxacin sequential therapy will be retreated with bismuth quadruple therapy for 10 days D1-D10: (esomeprazole 40mg bid + Dibismuth trioxide 120mg qid + metronidazole 500mg tid + tetracycline 500mg qid) for 10 days

Group (B) Patient who fail from bismuth quadruple therapy will be retreated with levofloxacin sequential therapy for 14days D1-D7: (esomeprazole 40mg bid + amoxicillin 1gm bid) for 7 days D8-D14: (esomeprazole 40mg bid + levofloxacin 250mg bid + metronidazole 500mg bid) for another 7 days

Outcome Measurement:

Primary End Point: Eradication rate in the second line according to intention to treat (ITT) and per-protocol (PP) analysis in the two treatment groups

ELIGIBILITY:
Inclusion Criteria:

1. H. pylori infected patients who failed from first line standard triple therapy with clarithromycin, amoxicillin, and a proton pump inhibitor were eligible in this study

Exclusion Criteria:

1. children and teenagers aged less than 20 years,
2. history of gastrectomy,
3. gastric malignancy, including adenocarcinoma and lymphoma,
4. previous allergic reaction to antibiotics (bismuth, metronidazole, levofloxacin, tetracycline) and PPI (esomeprazole),
5. contraindication to treatment drugs,
6. pregnant or lactating women,
7. severe concurrent disease, or
8. Unwilling to accept random assignment of subjects

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 560 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Eradication rate after second line eradication therapy according to ITT analysis | 6 weeks after completion of treatment
  The eradication status will be determined by urea breath test (UBT) at least 6 weeks after completion of the treatment. The delta value of UBT of 4 or less will be defined as negative and successful eradication.

SECONDARY OUTCOMES:
Adverse effects during eradication therapy | during treatment (2 weeks)
  adverse effects will be assessed by questionnaire
Long term eradication rate 1 year after eradication therapy | 1 year after treatment
  Long term eradication rates will be determined by UBT at 1 year after eradication therapy.
changes of gut microbiota before and after eradication therapy | 1 year
  Fecal DNA will be extracted and 16S rRNA sequencing will be done. The changes in the alpha and beta diversity and the compositions of gut microbiota before and after HP eradication will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Shiang Wu, Study Chair — National Taiwan University Hospital; Jyh-Ming Liou, Principal Investigator — National Taiwan University Hospital
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - National Taiwan University Hospital, Yunlin branch, Yunlin

IPD SHARING:
Plan to Share IPD: No
The investigators will not share the data.

REFERENCES:
- [Result] Liou JM, Chen CC, Chen MJ, Chen CC, Chang CY, Fang YJ, Lee JY, Hsu SJ, Luo JC, Chang WH, Hsu YC, Tseng CH, Tseng PH, Wang HP, Yang UC, Shun CT, Lin JT, Lee YC, Wu MS; Taiwan Helicobacter Consortium. Sequential versus triple therapy for the first-line treatment of Helicobacter pylori: a multicentre, open-label, randomised trial. Lancet. 2013 Jan 19;381(9862):205-13. doi: 10.1016/S0140-6736(12)61579-7. Epub 2012 Nov 16. PMID 23158886
- [Result] Liou JM, Chen CC, Chang CY, Chen MJ, Fang YJ, Lee JY, Chen CC, Hsu SJ, Hsu YC, Tseng CH, Tseng PH, Chang L, Chang WH, Wang HP, Shun CT, Wu JY, Lee YC, Lin JT, Wu MS; Taiwan Helicobacter Consortium. Efficacy of genotypic resistance-guided sequential therapy in the third-line treatment of refractory Helicobacter pylori infection: a multicentre clinical trial. J Antimicrob Chemother. 2013 Feb;68(2):450-6. doi: 10.1093/jac/dks407. Epub 2012 Oct 25. PMID 23099849
- [Result] Liou JM, Chen CC, Chen MJ, Chang CY, Fang YJ, Lee JY, Sheng WH, Wang HP, Wu MS, Lin JT. Empirical modified sequential therapy containing levofloxacin and high-dose esomeprazole in second-line therapy for Helicobacter pylori infection: a multicentre clinical trial. J Antimicrob Chemother. 2011 Aug;66(8):1847-52. doi: 10.1093/jac/dkr217. Epub 2011 May 31. PMID 21632579
- [Derived] Liou JM, Jiang XT, Chen CC, Luo JC, Bair MJ, Chen PY, Chou CK, Fang YJ, Chen MJ, Chen CC, Lee JY, Yang TH, Yu CC, Kuo CC, Chiu MC, Chen CY, Shun CT, Hu WH, Tsai MH, Hsu YC, Tseng CH, Chang CY, Lin JT, El-Omar EM, Wu MS; Taiwan Gastrointestinal Disease and Helicobacter Consortium. Second-line levofloxacin-based quadruple therapy versus bismuth-based quadruple therapy for Helicobacter pylori eradication and long-term changes to the gut microbiota and antibiotic resistome: a multicentre, open-label, randomised controlled trial. Lancet Gastroenterol Hepatol. 2023 Mar;8(3):228-241. doi: 10.1016/S2468-1253(22)00384-3. Epub 2022 Dec 19. PMID 36549320